CLINICAL TRIAL: NCT03291860
Title: Antimullerian Hormone as an Indicator fo Ovarian Response in Women Receiving Long GnRH Agonist Protocol in Intracytoplasmic Sperm Injection Cycles
Brief Title: Antimullerian Hormone as an Indicator for Ovarian Response
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Selim, Doctor, Ain Shams Maternity Hospital
Other Study IDs: Antimullerian hormone
Record Dates: First submitted 2017-09-18; First posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Ovum retrievum — assessment of oocytes collected by ovum retrievum to evaluate the discriminatory power of the antimullerian hormone in ICSI cycles

SUMMARY:
Anti Mullerian hormone (AMH) is gaining place as ovarian marker, chiefly in infertility assistance.

Investigators explored its correlation with oocytes retrieval after long GnRH agonist protocol for stimulation, in younger and older infertile population. Methods: This prospective analysis compiled data of 66 females, receiving ICSI treatment from April 2016 to October 2017. Serum FSH, LH, Estadiol, AMH and antral follicle count were assessed. Outcomes were measured as good (5 to 19 oocytes) and bad responders.

ELIGIBILITY:
Inclusion Criteria:

1. Age:20-40 years old
2. BMI:20-40kg/m
3. Normal baseline hormonal profile (on the 2nd day of the cycle)

   * FSH: 2.5-10.2mlU/ml
   * LH:1.9-12.5mlU/ml
   * Estradiol (E2): <50pg/ml
4. No Endometriosis by laparoscopy
5. No prior ovarian surgery; overectomy, ovariectomy or oophrectomy
6. Female subjects who have at least 1 wash-out cycle (defined as greater than or equal to 30 days since the last dose of clomiphene citrate or gonadotrophin treatment) since the last ART cycle and/or clomiphene citrate or gonadotrophin treatment prior to starting gonadotrophin releasing hormone (GnRH) agonist therapy

Exclusion Criteria:

* 1. Age: <20 or >40 years old 2. BMI: <20 or >40kg/m 3. Female subjects with any contraindication for pregnancy. 4. Female subjects with history of tumors of the hypothalamus & pituitary gland.

  5. Female subjects with history of ovarian, uterine or mammary cancer. 6. Female subjects with history of hypersensitivity to the active substance of the medications used for ovarian stimulation.

  7. Abnormal baseline hormonal profile 8. Endometriosis by laparoscopy 9. Previous ovarian surgery; overectomy, ovariectomy or oophrectomy 10. Female subjects with abnormal gynecological bleeding of unknown etiology

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Sixty six women undergoing ICSI were enrolled in and a written informed consent was obtained from each participant
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2017-11-10 (Estimated); Primary Completion 2018-09-10 (Estimated); Study Completion 2018-10-10 (Estimated)

PRIMARY OUTCOMES:
Difference between AMH levels between good and poor responders in young patients receiving long GnRH agonist protocol for ICSI. | 1 month (1 cycle)
  Measurement of AMH level in patients undergoing controlled ovarian stimulation prior to ICSI using long GnRH agonist protocol. Level will be compared between good and poor responders.